CLINICAL TRIAL: NCT02888665
Title: A Trial of Pembrolizumab in Combination With Doxorubicin as Treatment for Patients With Advanced Sarcomas
Brief Title: Pembrolizumab and Doxorubicin Hydrochloride in Treating Patients With Sarcoma That is Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Seth Pollack, Steven T. Rosen, MD, Professor of Cancer Biology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9624; NCI-2016-01286 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9624 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG9216017 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pembrolizumab, doxorubicin hydrochloride) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and doxorubicin hydrochloride IV over 1-3 hours on day 1 of courses 2-7 only. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I/II trial studies the side effects and best dose of doxorubicin hydrochloride when given together with pembrolizumab and to see how well they work in treating patients with sarcoma that have spread to other parts of the body or that cannot be removed by surgery. Drugs used in chemotherapy, such as doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving doxorubicin hydrochloride together with pembrolizumab may work better in treating patients with sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of the combination of pembrolizumab and doxorubicin hydrochloride (doxorubicin) in patients with advanced soft tissue sarcoma (STS).

II. To assess the clinical response rate of advanced soft tissue sarcoma (STS) patients receiving the combination of pembrolizumab and doxorubicin.

SECONDARY OBJECTIVES:

I. To explore the clinical activity of pembrolizumab in subjects with advanced STS with respect to time to response.

II. To explore the clinical activity of pembrolizumab in subjects with advanced STS with respect to duration of response.

III. To explore the clinical activity of pembrolizumab in subjects with advanced STS with respect to progression-free survival (PFS).

IV. To explore the clinical activity of pembrolizumab in subjects with advanced STS with respect to overall survival.

TERTIARY OBJECTIVES:

I. To compare response rates between patients with high levels of PD-L1 expression with those who have PD-L1 absent.

OUTLINE: This is a phase I, dose-escalation study of doxorubicin hydrochloride followed by a phase II study.

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and doxorubicin hydrochloride IV over 1-3 hours on day 1 of courses 2-7 only. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Have metastatic or unresectable sarcoma
* Have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500/mcL (within 10 days of treatment initiation)
* Platelets >= 100,000/mcL (within 10 days of treatment initiation)
* Hemoglobin >= 9 g/dL (within 10 days of treatment initiation) or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (within 10 days of treatment initiation)
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (within 10 days of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases (within 10 days of treatment initiation)
* Albumin >= 2.5 mg/dL (within 10 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 10 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (within 10 days of treatment initiation)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Ejection fraction > 45% by either multi-gated acquisition scan (MUGA) scan or echocardiogram

Exclusion Criteria:

* Has prior treatment using an anthracycline
* Has one of the following sarcoma subtypes where combining anthracyclines with other chemotherapies is established as the standard of care: osteosarcoma, Ewings sarcoma, embryonal rhabdomyosarcoma, alveolar rhabdomyosarcoma
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-programed death receptor 1 (PD-1), anti-PD-L1, anti-program death receptor ligand 2 (PD-L2) agent or anti-CTLA4
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Pollack, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Pollack SM, Redman MW, Baker KK, Wagner MJ, Schroeder BA, Loggers ET, Trieselmann K, Copeland VC, Zhang S, Black G, McDonnell S, Gregory J, Johnson R, Moore R, Jones RL, Cranmer LD. Assessment of Doxorubicin and Pembrolizumab in Patients With Advanced Anthracycline-Naive Sarcoma: A Phase 1/2 Nonrandomized Clinical Trial. JAMA Oncol. 2020 Nov 1;6(11):1778-1782. doi: 10.1001/jamaoncol.2020.3689. PMID 32910151

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1, Part 1: Subjects received 45 mg/m2 doxorubicin plus 200 mg flat dose of pembrolizumab.
- Phase 1, Part 2: Subjects received 75 mg/m2 doxorubicin + 200 mg flat dose of pembrolizumab.
- Phase 2: Subjects received 75 mg/m2 doxorubicin + 200 mg flat dose pembrolizumab.
Period: Overall Study
Arm/Group | Phase 1, Part 1 | Phase 1, Part 2 | Phase 2
Started | 3 | 3 | 31
Completed | 3 | 3 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1, Part 1 | Phase 1, Part 2 | Phase 2 | Total
Number analyzed (Participants) | 3 | 3 | 31 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 23 | 27
  >=65 years | 1 | 1 | 8 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 14 | 15
  Male | 3 | 2 | 17 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 4 | 5
  Not Hispanic or Latino | 3 | 2 | 26 | 31
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 3 | 2 | 22 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Doxorubicin Hydrochloride Plus Pembrolizumab According to the National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) Version 4.0 (Phase I)
Description: Defined as a dose limiting toxicity (DLT) in less than 2 of 6 subjects. Only Phase 1 subjects will be evaluated for MTD.
Time Frame: Up to 42 days (6 weeks)
Population: Only Phase 1 subjects were evaluated for a Maximum Tolerated Dose (MTD) based off of Dose-Limiting Toxicities experienced per subject as defined in the protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Cohort 1: Subjects received 45 mg/m2 of doxorubicin plus 200 mg flat dose of pembrolizumab.
- Phase 1 Cohort 2: Subjects received 75 mg/m2 of doxorubicin plus 200 mg flat dose of pembrolizumab.
Arm/Group | Phase 1 Cohort 1 | Phase 1 Cohort 2
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

2. Primary Outcome: Objective Response Rate (ORR) (Phase II)
Description: Evaluated per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT. Complete Response (CR) is a complete elimination of the tumor; Partial Response (PR) is 30% reduction. If a subject experienced a PR, this was required to be confirmed with a second scan at the next appropriate cycle.
Time Frame: Up to 2 years
Population: Only Phase 2 subjects were evaluated for this outcome as Phase 1 subjects were only included in the protocol for safety evaluation.
Measure: Number; unit: percent of participants
Groups:
- Phase 2: Treatment (Pembrolizumab, Doxorubicin Hydrochloride): Patients receive pembrolizumab IV over 30 minutes on day 1 and doxorubicin hydrochloride IV over 1-3 hours on day 1 of courses 2-7 only. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Doxorubicin Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
Arm/Group | Phase 2: Treatment (Pembrolizumab, Doxorubicin Hydrochloride)
Number analyzed (Participants) | 31
percent of participants | 13
Statistical Analysis 1: Comparison: Phase 2: Treatment (Pembrolizumab, Doxorubicin Hydrochloride); The primary objective of the phase II design compared ORR with historical rates (Judson et al. Lancet Onc., 2014). A 2-stage design with null hypothesis of 15% using a 1-sided 0.05 α level test has 85% power to detect an increase to 35%. This required up to 35 patients. After 2 responses in stage 1 (20 pts), the study moved to stage 2 (15 pts). If 10 responses were seen (29%), this would have ruled out an ORR of 15%. The study was closed when it became clear we would not meet this benchmark; Test type: Other; see above. target ORR was not met; see above — see above. target ORR was not met; see above. target ORR was not met

3. Secondary Outcome: Duration of Response
Description: Duration of response is the mean time to progression for all subjects who responded.
Time Frame: Up to 2 years
Population: Only 5 appropriate subjects had partial responses for evaluation.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Treatment (Pembrolizumab, Doxorubicin Hydrochloride)
Number analyzed (Participants) | 5
Days | 247 (180)

4. Secondary Outcome: Median Progression-free Survival (PFS)
Description: The Kaplan-Meier method will be used to estimate median PFS.
Time Frame: Up to 2 years
Population: This combined the phase I and phase II populations as we had intended for this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Doxorubicin Hydrochloride)
Number analyzed (Participants) | 37
months | 8.1 [7.6 to 10.8]

5. Secondary Outcome: Overall Survival (OS)
Description: The Kaplan-Meier method will be used to estimate median OS.
Time Frame: Up to 2 years
Population: This combined the phase I and phase II populations as we had intended for this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Doxorubicin Hydrochloride)
Number analyzed (Participants) | 37
months | 27.6 [18.7 to NA] — At the time of the final analysis, the upper limit had not yet been reached.

6. Secondary Outcome: Time to Response
Description: Average time to response
Time Frame: Up to 2 years
Population: Only 5 appropriate subjects had partial responses for evaluation.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Treatment (Pembrolizumab, Doxorubicin Hydrochloride)
Number analyzed (Participants) | 5
Days | 152.2 (65)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected beginning from date of consent to 30 days post discontinuation of study treatment. (Up to 2 years of therapy with 1 cycle equaling 21 days)
Groups:
- Phase 1 Cohort 1: Subjects received 45 mg/m2 doxorubicin plus 200 mg flat dose of pembrolizumab.
- Phase 1 Cohort 2: Subjects received 75 mg/m2 doxorubicin plus 200 mg flat dose of pembrolizumab.
- Phase 2: Subjects received 75 mg/m2 doxorubicin plus 200 mg flat dose pembrolizumab.
Arm/Group | Phase 1 Cohort 1 | Phase 1 Cohort 2 | Phase 2
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/3 | 15/31
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 13/31
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1 (N=3) | Phase 1 Cohort 2 (N=3) | Phase 2 (N=31)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Elevated troponin (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Investigations) | 0 (0) | 0 (0) | 1 (1)
Atypical Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Postprandial Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Partial Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Mid-esophageal erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Denuded mucosa (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsions (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vasovalgal reaction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Right lower lobe infiltrate (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary infarct (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor thrombus (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal thrush (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Kidney Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1 (N=3) | Phase 1 Cohort 2 (N=3) | Phase 2 (N=31)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 27 (37)
Fatigue (General disorders) | 1 (1) | 3 (3) | 21 (26)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 2 (3) | 14 (19)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 12 (16)
Fever (General disorders) | 1 (1) | 2 (2) | 13 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 11 (11)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 14 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 11 (12)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 9 (12)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (3) | 12 (16)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (3) | 9 (9)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 12 (16)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 8 (9)
Neutrophil Count Decreased (Investigations) | 0 (0) | 2 (3) | 7 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 9 (11)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 7 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 7 (9)
Dry Eye (Eye disorders) | 1 (1) | 3 (3) | 5 (5)
Weight Loss (Investigations) | 0 (0) | 1 (1) | 7 (18)
Pain (General disorders) | 0 (0) | 1 (3) | 7 (7)
Edema Limbs (General disorders) | 1 (1) | 1 (1) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 7 (13)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 7 (7)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 8 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 7 (7)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 8 (11)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1) | 8 (11)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 8 (8)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 5 (7)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 6 (8)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (4)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 5 (7)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 8 (11)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (7)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 4 (4)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 4 (4)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (5)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (6)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0) | 4 (4)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 3 (4)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0) | 3 (4)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (9)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 3 (3)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (2) | 2 (2)
Alanine aminotransferase increase (Investigations) | 0 (0) | 0 (0) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 3 (4)
Sore throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Right Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (4)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (4)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4)
Eye Pain (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Hemoptysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Bilateral anterior uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion Related Reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Left Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Squamous Cell Carcinoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Restless Legs (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Bump on Elbow (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tinea Pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Seborrheic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Small Bump on Right Shoulder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Sensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain at Port Site (General disorders) | 1 (1) | 0 (0) | 0 (0)
Delayed word recall (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Right Upper Extremity Numbness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Left Upper Extremity Numbness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Rib Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Incomplete Right Bundle Branch Lock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Palatal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shoulder Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sebaceous cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal Discharge (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT02888665/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT02888665/ICF_001.pdf